CLINICAL TRIAL: NCT03842969
Title: An Open-Label Extension Study to Evaluate the Long-Term Safety and Tolerability of Intrathecally Administered RO7234292 (RG6042) in Patients With Huntington's Disease
Brief Title: An Open-Label Extension Study to Evaluate Long-Term Safety and Tolerability of RO7234292 (RG6042) in Huntington's Disease Participants Who Participated in Prior Roche and Genentech Sponsored Studies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BN40955; 2018-003898-94 (EudraCT Number)
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Results first posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — tominersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RO7234292 (RG6042) Q8W (Experimental): Participants who received open-label RO7234292 Q4W in a preceding study or who received RO7234292 Q4W in this study may be randomly allocated to receive RO7234292 Q8W. Participants who previously received open-label of RO7234292 Q8W in a preceding study or are currently receiving RO7234292 Q8W in this study will receive RO7234292 Q8W. Participants who previously received placebo, or did not previously receive treatment with RO7234292 or received short-term treatment with a treatment-free follow-up period may be randomly allocated to receive RO7234292 Q8W. Participants who previously received blinded placebo Q8W may receive RO7234292 Q8W. Participants who received blinded RO7234292 Q8W will receive open-label RO7234929 Q8W. Participants who received blinded placebo Q8W may receive RO7234292 Q8W. Participants who received blinded RO7234292 Q4W or blinded placebo Q4W may be randomly allocated to receive open-label of RO7234292 Q8W.
  Interventions: Drug: RO7234292 (RG6042)
- RO7234292 (RG6042) Q16W (Experimental): Participants who previously received open-label RO7234292 Q4W in a preceding study or who received RO7234292 Q4W in this study may be randomly allocated to receive RO7234292 Q16W. Participants who previously received placebo in a preceding study or did not previously receive treatment with RO7234292 or received short-term treatment with a treatment-free follow-up period may be randomly allocated to receive RO7234292 Q16W. Participants who previously received blinded placebo Q8W will receive RO7234292 Q8W. Participants who previously received blinded RO7234292 Q16W will receive open-label RO7234292 Q16W. Participants who received blinded RO7234292 Q4W or blinded placebo Q4W may be randomly allocated to receive open-label of RO7234292 Q16W. Participants who previously received open-label RO7234292 Q16W will receive open-label RO7234292 Q16W.
  Interventions: Drug: RO7234292 (RG6042)

INTERVENTIONS:
Drug: RO7234292 (RG6042) — Intrathecal injection
  Other Names: Tominersen

SUMMARY:
This study will evaluate the long-term safety and tolerability of RO7234292 (RG6042) in participants who have completed other F. Hoffmann-La Roche, Ltd.-sponsored and/or Genentech-sponsored studies in the Huntington's disease (HD) in the development program for RG6042.

DETAILED DESCRIPTION:
Entry into the study should occur at the time the participant completes participation in one of the preceding studies. Upon completion of the inclusion visit, eligible participants will receive either RO7234292 (RG6042) every 8 weeks (Q8W) or RO7234292 (RG6042) every 16 weeks (Q16W) by the bolus intrathecal injection.

ELIGIBILITY:
Inclusion Criteria:

* Prior enrollment in a Roche-sponsored or Genentech-sponsored study in HD for the RO7234292 (RG6042) development program that made provision for entry into an OLE study
* For women of childbearing potential: agreement to remain abstinent or use contraceptive measures
* For men: agreement to remain abstinent or use a condom, and agreement to refrain from donating sperm
* Patients who were screened and eligible for the placebo-controlled Phase III Study BN40423 but could not be randomized prior to the close of Study BN40423 enrollment due to challenges relating to the COVID-19 pandemic

Inclusion criteria of patients who were screened and eligible for the placebo-controlled Phase III Study BN40423 but could not be randomized prior to the close of Study BN40423 enrollment due to challenges relating to the COVID-19 pandemic:

* Manifest HD diagnosis, defined as a DCL score of 4
* Independence Scale (IS) score >=70
* Genetically confirmed disease by direct DNA testing with a CAP score >400
* Clinical assessment to ensure individual has intact functional independence at baseline to maintain self-care and core activities of daily living (ADLs).

Exclusion Criteria:

* Withdrawal of consent from the preceding study
* Permanent discontinuation of RO7234292 (RG6042) for any drug-related safety concern during the preceding study or meeting of any study treatment discontinuation criteria specified in the preceding study at the time of enrollment into this study
* An ongoing, unresolved, clinically significant medical problem that in the judgment of the investigator would make it unsafe for the patient to participate in this study
* Antiplatelet or anticoagulant therapy within 14 days prior to inclusion or anticipated use during the study, including, but not limited to, aspirin, clopidogrel, dipyridamole, warfarin, dabigatran, rivaroxaban, and apixaban
* History of bleeding diathesis or coagulopathy
* Platelet count less than the lower limit of normal
* Concurrent participation in any therapeutic clinical trial
* Study treatment (RO7234292/RG6042) is commercially marketed in the patient's country for the patient-specific disease and is accessible to the patient
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 5 months after the final dose of study drug

Exclusion criteria of patients who were screened and eligible for the placebo-controlled Phase III Study BN40423 but could not be randomized prior to the close of Study BN40423 enrollment due to challenges relation to the COVID-19 pandemic:

* Any serious medical condition or clinically significant laboratory, or vital sign abnormality or claustrophobia at screening that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 5 months after the final dose of study drug

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- United States (14):
  - Uab Medicine, Birmingham, Alabama
  - University of California San Diego, La Jolla, California
  - Stanford Univ Medical Center, Palo Alto, California
  - SC3 Research Group, Inc, Pasadena, California
  - CenExel Rocky Mountain Clinical Research, LLC, Englewood, Colorado
  - Georgetown University; Research Division, Psychiatry, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Dent Neurological Institute, Amherst, New York
  - Columbia University, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Health Science Center at Houston; McGovern Medical School, Houston, Texas
- Uniklinik fuer Neurologie, Medizinische Universitaet Innsbruck; Department fuer Neurologie, Innsbruck, Austria
- Canada (4):
  - University of British Columbia Hospital; Division of Neurology, Vancouver, British Columbia
  - Centre for Movement Disorders, North YORK, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Centre Hospitalier de l?Université de Montréal (CHUM), Montreal, Quebec
- Germany (3):
  - Charité - Universitätsmed. Berlin, Klinik für Psychiatrie und Psychotherapie; Abt. Neuropsychiatrie, Berlin
  - St. Josef-Hospital, Neurologische Klinik der Ruhr-Uni; Huntington-Center NRW, Abt. Neurodegeneration, Bochum
  - Universitätsklinikum Ulm; Klinik für Neurologie, Ulm
- Italy (2):
  - IRCCS Casa Sollievo Della Sofferenza; Unità Ricerca e Cura Huntington e Malattie Rare, San Giovanni Rotondo (FG), Apulia
  - Fondazione IRCCS Istituto Neurologico Carlo Besta; U.O.C. Genetica Medica-Neurogenetica, Milan, Lombardy
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - LUMC, Leiden
- Spain (7):
  - Hospital Universitario de Badajoz; Servicio de Neurología, Badajoz
  - Hospital Clinic Servicio de Neurologia, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Neurologia, Barcelona
  - Hospital Universitario de Burgos. Servicio de Neurología, Burgos
  - Hospital Ramon y Cajal; Servicio de Neurologia, Madrid
  - Fundacion Jimenez Diaz; Servicio de Neurología, Madrid
  - Hospital Universitario Virgen Macarena; Servicio de Neurologia, Seville
- United Kingdom (5):
  - Birmingham and Solihull Mental Health Foundation Trust; Institute of Clinical Sciences, Birmingham
  - Cambridge Centre for Brain Repair; Department of Clinical Nuerosciences, Addenbrookes Hospital, Cambridge
  - University Hospital of Wales; Division of Psychological Medicine and Clinical Neurosciences, Cardiff
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London
  - Central Manchester University Hospitals NHS Foundation Trust; Manchester Centre for Genomic Medicine, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consists of Period 1 and 2. All participants (17) in the Q4W arm stopped Q4W dosing (Period 1) and 15 participants continued into the two Arms of Period 2. Due to the statistical outputs available, Period 1 and 2 are reported as Milestones below. None of the participants completed the study.
Pre-assignment Details: Periods 1 and 2 are sequential. 15 from 17 participants from Period 1 Q4W were re-randomized to receive Tominersen 120 mg Q8W or Q16W in Period 2 randomly and blinded.
  .
Groups:
- Tominersen 120mg Q4W: Participants received open-label RO7234292 Q4W in this Arm
- Tominersen 120mg Q8W: Participants received open-label RO7234292 Q8W in this Arm
- Tominersen 120mg Q16W: Participants received open-label RO7234292 Q16W in this Arm
Period: Overall Study
Arm/Group | Tominersen 120mg Q4W | Tominersen 120mg Q8W | Tominersen 120mg Q16W
Started | 17 | 138 | 81
Period 1 (Period 1 has only 1 arm with 17 participants of which 15 were transferred to two Arms of Period 2 (8 and 7 participants, see below)) | 17 | 0 | 0
Period 2 (Period 2 has 2 arms: Tominersen 120mg Q8W (8 participants from Period 1 and 138 new participants enrolled) and Tominersen 120mg Q16W (7 participants from Period 1 and 81 new enrolled). There were no participants in arm Tominersen 120mg Q4W.) | 0 (8 and 7 Participants from Arm Tominersen 120mg Q4W (Period 1) joined newly enrolled 138 participants in this Arm of Period 2.) | 146 (8 Participants from Arm Tominersen 120mg Q4W (Period 1) joined newly enrolled 138 participants in this Arm of Period 2.) | 88 (7 Participants from Arm Tominersen 120mg Q4W (Period 2) joined newly enrolled 81 participants in this Arm of Period 2)
Completed (None of the participants completed the study) | 0 | 0 | 0
Not Completed | 17 | 138 | 81
Not completed — Participant declined follow-up visit | 0 | 1 | 0
Not completed — Sponsor's decision | 12 | 99 | 61
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Death | 1 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 30 | 18
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Physician Decision | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: In Period 1 Milestone, 17 participants received 120 mg Tominersen Q4W Arm.
  In the Milestone Period 2, 138 and 81 participants received 120 mg Tominersen Q8W and Q16W respectively, with 15 participants from the In Period 1 Milestone Arm. 8 and 7 participants from Period 1 joined the two arms of Period 2. Period 2 did not have the arm Tominersen 120mg Q4W.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tominersen 120mg Q4W | Tominersen 120mg Q8W | Tominersen 120mg Q16W | Total
Number analyzed (Participants) | 17 | 138 | 81 | 236
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population description: In the Milestone Period 2, 146 and 88 participants received 120 mg Tominersen Q8W and Q16W respectively, with 15 participants from the In Period 1 Milestone Arm. There is no data to report separately for Milestone Periods 1 and 2 as no such statistical analyses were performed without 15 participants from the Milestone Period 1 in Milestone Period 2. Population: After Period 1, 15 patients continued to Period 2 with re-randomization
  Years
    Period 1: number analyzed (Participants) | 17 | 0 | 0 | 17
    Period 1 | 50.4 (8.9) |  |  | 50.4 (8.9)
    Period 2: number analyzed (Participants) | 0 | 138 | 81 | 219
    Period 2 |  | 47.9 (9.8) | 48.4 (11.2) | 48.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population Description: In the Milestone Period 2, 146 and 88 participants received 120 mg Tominersen Q8W and Q16W respectively, with 15 participants from the In Period 1 Milestone Arm. There is no data to report separately for Milestone Periods 1 and 2 as no such statistical analyses were performed without 15 participants from the Milestone Period 1 in Milestone Period 2. Population: After Period 1, 15 patients continued to Period 2 with re-randomization
  Participants
    Period 1: number analyzed (Participants) | 17 | 0 | 0 | 17
    Period 1: Female | 6 | 0 | 0 | 6
    Period 1: Male | 11 | 0 | 0 | 11
    Period 2: number analyzed (Participants) | 0 | 138 | 81 | 219
    Period 2: Female | 0 | 71 | 37 | 108
    Period 2: Male | 0 | 67 | 44 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population Description: In the Milestone Period 2, 146 and 88 participants received 120 mg Tominersen Q8W and Q16W respectively, with 15 participants from the In Period 1 Milestone Arm. There is no data to report separately for Milestone Periods 1 and 2 as no such statistical analyses were performed without 15 participants from the Milestone Period 1 in Milestone Period 2. Population: After Period 1, 15 patients continued to Period 2 with re-randomization
  Participants
    Period 1: number analyzed (Participants) | 17 | 0 | 0 | 17
    Period 1: Hispanic or Latino | 0 | 0 | 0 | 0
    Period 1: Not Hispanic or Latino | 17 | 0 | 0 | 17
    Period 1: Unknown or Not Reported | 0 | 0 | 0 | 0
    Period 2: number analyzed (Participants) | 0 | 138 | 81 | 219
    Period 2: Hispanic or Latino | 0 | 13 | 7 | 20
    Period 2: Not Hispanic or Latino | 0 | 125 | 74 | 199
    Period 2: Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population Description: In the Milestone Period 2, 146 and 88 participants received 120 mg Tominersen Q8W and Q16W respectively, with 15 participants from the In Period 1 Milestone Arm. There is no data to report separately for Milestone Periods 1 and 2 as no such statistical analyses were performed without 15 participants from the Milestone Period 1 in Milestone Period 2. Population: After Period 1, 15 patients continued to Period 2 with re-randomization
  Participants
    Period 1: number analyzed (Participants) | 17 | 0 | 0 | 17
    Period 1: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Period 1: Asian | 0 | 0 | 0 | 0
    Period 1: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Period 1: Black or African American | 0 | 0 | 0 | 0
    Period 1: White | 17 | 0 | 0 | 17
    Period 1: More than one race | 0 | 0 | 0 | 0
    Period 1: Unknown or Not Reported | 0 | 0 | 0 | 0
    Period 2: number analyzed (Participants) | 0 | 138 | 81 | 219
    Period 2: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Period 2: Asian | 0 | 2 | 1 | 3
    Period 2: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Period 2: Black or African American | 0 | 2 | 0 | 2
    Period 2: White | 0 | 132 | 76 | 208
    Period 2: More than one race | 0 | 1 | 1 | 2
    Period 2: Unknown or Not Reported | 0 | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events
Description: The reported are the treatment-emergent AEs with an onset date up to 5 months after last study drug intake.
Time Frame: Up to Approximately 3 Years
Population: Safety Population
Measure: Number; unit: Percentage of Participants
Groups:
- Tominersen 120 mg Q8W: Participants received open-label RO7234292 Q8W in this Arm
- Tominersen 120 mg Q16W: Participants received open-label RO7234292 Q16W in this Arm
Arm/Group | Tominersen 120mg Q4W | Tominersen 120 mg Q8W | Tominersen 120 mg Q16W
Number analyzed (Participants) | 14 | 143 | 88
Percentage of Participants | 71.4 | 83.9 | 81.8

2. Primary Outcome: Number of Participants With Suicidal Ideation, Suicidal Behavior, and Self-Injurious Behavior Without Suicidal Intent Based on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is to assess suicidal ideation and behavior. 4 constructs measured: severity of ideation, intensity of ideation, behavior, and lethality of actual suicide attempts. Yes/No data collected for 10 categories, composite endpoints based on the categories are followed over time to monitor safety. Composite endpoint of suicidal ideation (1-5), n and (%) are the number and % of who experience any of the five suicidal ideation events at least once after receiving the first dose of study medication. Composite endpoint of suicidal behavior (6-10), n and (%) are the number and percent of patients who experience any 1of 5 suicidal behavior events at least 1 after receiving the 5 dose of study medication. Composite endpoint of suicidal ideation or behavior (1-10), n and (%) are the number and % of patients who experience any 1 the 10 suicidal ideation or behavior events at least once after receiving the first dose of study medication.
Time Frame: Up to approximately 3 Years
Population: Safety Population. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) are included. All other data were not evaluable due to participants' discontinuation
Measure: Number; unit: Number of participants
Arm/Group | Tominersen 120mg Q4W | Tominersen 120 mg Q8W | Tominersen 120mg Q16W
Number analyzed (Participants) | 14 | 143 | 88
Number of participants
  Suicidal Ideation (1-5) -Wish to Be Dead | 1 | 16 | 3
  Suicidal Ideation (1-5) -Non-specific Active Suicidal Thoughts | 0 | 9 | 1
  Suicidal Ideation (1-5) -Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act | 0 | 7 | 1
  Suicidal Ideation (1-5) -Active Suicidal Ideation with Intent to Act, without Specific Plan | 0 | 3 | 1
  Suicidal Ideation (1-5) -Active Suicidal Ideation with Specific Plan and Intent | 0 | 2 | 0
  Suicidal Behavior (6-10) -Preparatory Acts or Behavior | 0 | 1 | 0
  Suicidal Behavior (6-10) -Aborted Attempt | 0 | 0 | 0
  Suicidal Behavior (6-10) -Interrupted Attempt | 0 | 1 | 0
  Suicidal Behavior (6-10) -Non-fatal Suicide Attempt | 0 | 2 | 0
  Suicidal Behavior (6-10) -Completed Suicide | 0 | 0 | 0
  Suicidal Ideation or Behavior (1-10) | 1 | 16 | 3
  Self-injurious Behavior without Suicidal Intent | 0 | 1 | 0
  Treatment-Emergent Suicidal Ideation: number analyzed (Participants) | 14 | 140 | 81
  Treatment-Emergent Suicidal Ideation | 0 | 14 | 2
  Treatment-Emergent Serious Suicidal Ideation: number analyzed (Participants) | 14 | 140 | 80
  Treatment-Emergent Serious Suicidal Ideation | 0 | 3 | 1
  Emergence of Serious Suicidal Ideation: number analyzed (Participants) | 13 | 135 | 80
  Emergence of Serious Suicidal Ideation | 0 | 2 | 1
  Emergence of Suicidal Behavior: number analyzed (Participants) | 14 | 140 | 80
  Emergence of Suicidal Behavior | 0 | 3 | 0

3. Primary Outcome: Change From Baseline in Cognition, Using Montreal Cognitive Assessment (MoCA)
Description: MoCA contains a series of basic assessments, including attention and visuospatial tasks. The total score ranges from 0-30, where lower scores indicate greater impairment.
  MOCA01-Total scores are reported. The data presented are absolute scores for baseline and change from baseline for post-baseline assessments.
  All Arms except Tominersen 120mg Q4W (Period 1) belong to the Milestone Period 2.
Time Frame: Up to Approximately 3 Years
Population: Safety Population. Data evaluable participants were reported, all other data are not available. Only those participants who contributed and whose data were analyzed for data are reported in the table.
Measure: Mean (Standard Deviation); unit: Score of a Scale
Groups:
- Tominersen 120mg Q4W (Period 1): Period 1 Tominersen 120mg Q4W Participants received open-label RO7234292 Q4W in this Period 1
- Tominersen 120mg Q8W (Prior Q4w): Participants received open-label RO7234292 Q8W after having received Q4W treatment previously
- Tominersen 120mg Q8W (No Loading): Participants received open-label RO7234292 Q8W without prior treatment with RO7234292
- Tominersen 120mg Q8W (With Loading): Participants received open-label RO7234292 Q8W with prior treatment with RO7234292 Q8W
- Tominersen 120mg Q8W (Prior BP40410): Participants received open-label RO7234292 Q8W with prior treatment with RO7234292 Q4W in study BP40410
- Tominersen 120mg Q16W (Prior Q4W): Participants received open-label RO7234292 Q16W after having received Q4W treatment previously
- Tominersen 120mg Q16W (No Loading): Participants received open-label RO7234292 Q16W without prior treatment with RO7234292
- Tominersen 120mg Q16W (Prior BP40410): Participants received open-label RO7234292 Q16W with prior treatment with RO7234292 Q4W in study BP40410
Arm/Group | Tominersen 120mg Q4W (Period 1) | Tominersen 120mg Q8W (Prior Q4w) | Tominersen 120mg Q8W (No Loading) | Tominersen 120mg Q8W (With Loading) | Tominersen 120mg Q8W (Prior BP40410) | Tominersen 120mg Q16W (Prior Q4W) | Tominersen 120mg Q16W (No Loading) | Tominersen 120mg Q16W (Prior BP40410)
Number analyzed (Participants) | 14 | 25 | 72 | 43 | 3 | 24 | 60 | 4
Score of a Scale
  MOCA01-Total Baseline: number analyzed (Participants) | 14 | 25 | 66 | 42 | 3 | 23 | 58 | 4
  MOCA01-Total Baseline | 24.50 (3.98) | 25.08 (3.49) | 24.92 (3.47) | 24.62 (4.44) | 25.33 (1.53) | 23.43 (4.49) | 24.03 (3.88) | 19.75 (4.35)
  MOCA01-Total Week 17: number analyzed (Participants) | 1 | 24 | 63 | 36 | 3 | 21 | 53 | 4
  MOCA01-Total Week 17 | -4.00 (NA) — No data available in the range | 0.46 (2.19) | 0.16 (2.58) | 0.19 (2.56) | -1.00 (1.00) | -0.57 (2.01) | -0.17 (2.79) | 3.25 (2.36)
  MOCA01-Total Week 25: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MOCA01-Total Week 25 | 3.00 (NA) — No data available in the range |  |  |  |  |  |  |
  MOCA01-Total Week 33: number analyzed (Participants) | 1 | 19 | 58 | 34 | 3 | 21 | 47 | 4
  MOCA01-Total Week 33 | 3.00 (NA) — No data available in the range | 0.16 (1.74) | 0.28 (2.61) | 0.35 (1.76) | 0.67 (2.08) | -0.90 (2.76) | 0.32 (2.44) | 2.25 (2.22)
  MOCA01-Total Week 49: number analyzed (Participants) | 0 | 24 | 57 | 36 | 3 | 20 | 53 | 3
  MOCA01-Total Week 49 |  | 0.33 (2.33) | -0.39 (2.83) | -0.08 (2.26) | -0.67 (3.06) | -0.40 (2.68) | -0.13 (2.53) | 3.00 (3.46)
  MOCA01-Total Week 65: number analyzed (Participants) | 0 | 23 | 53 | 40 | 1 | 21 | 48 | 2
  MOCA01-Total Week 65 |  | -0.09 (2.09) | -0.08 (2.56) | -0.08 (1.91) | -5.00 (NA) — No data available in the range | -0.43 (2.86) | 0.27 (2.85) | 0.50 (3.54)
  MOCA01-Total Week 81: number analyzed (Participants) | 0 | 22 | 45 | 35 | 1 | 20 | 41 | 2
  MOCA01-Total Week 81 |  | 0.59 (1.30) | -0.38 (3.31) | -0.09 (1.95) | -2.00 (NA) — No data available in the range | 0.25 (2.57) | -0.24 (2.90) | 0.50 (3.54)
  MOCA01-Total Week 97: number analyzed (Participants) | 0 | 19 | 30 | 31 | 0 | 17 | 24 | 0
  MOCA01-Total Week 97 |  | -0.47 (2.06) | -0.97 (3.12) | 0.45 (2.20) |  | 0.24 (2.46) | -0.46 (3.01) |
  MOCA01-Total Week 113: number analyzed (Participants) | 0 | 17 | 22 | 30 | 0 | 16 | 11 | 0
  MOCA01-Total Week 113 |  | 0.18 (1.94) | -0.36 (2.65) | 0.10 (2.62) |  | 0.19 (2.51) | 0.36 (3.01) |
  MOCA01-Total Week 129: number analyzed (Participants) | 0 | 12 | 14 | 20 | 0 | 9 | 5 | 0
  MOCA01-Total Week 129 |  | -0.75 (1.22) | -0.50 (1.95) | -0.15 (3.48) |  | -0.11 (1.90) | 2.20 (3.19) |
  MOCA01-Total Week 145: number analyzed (Participants) | 0 | 3 | 0 | 6 | 0 | 1 | 0 | 0
  MOCA01-Total Week 145 |  | 0.33 (1.53) |  | -4.83 (5.91) |  | 0.00 (NA) — No data available in the range |  |

ADVERSE EVENTS:
Time Frame: Up to Approx. 3 Years
Arm/Group | Tominersen 120mg Q4W | Tominersen 120 mg Q8W | Tominersen 120 mg Q16W
All-Cause Mortality (participants affected / at risk) | 1/14 | 0/143 | 1/88
Serious Adverse Events (participants affected / at risk) | 1/14 | 17/143 | 9/88
Other Adverse Events (participants affected / at risk) | 12/14 | 99/143 | 56/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tominersen 120mg Q4W (N=14) | Tominersen 120 mg Q8W (N=143) | Tominersen 120 mg Q16W (N=88)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Arachnoiditis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Chorea (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Dissociative disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (3)
Suicidal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Euthanasia (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tominersen 120mg Q4W (N=14) | Tominersen 120 mg Q8W (N=143) | Tominersen 120 mg Q16W (N=88)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 9 (9) | 5 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 5 (5) | 4 (5)
Gait disturbance (General disorders) | 0 (0) | 3 (4) | 5 (5)
Oedema peripheral (General disorders) | 1 (1) | 2 (3) | 0 (0)
Injection site infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 13 (15) | 3 (3)
Onychomycosis (Infections and infestations) | 1 (1) | 1 (1) | 1 (2)
Tooth infection (Infections and infestations) | 1 (1) | 2 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 5 (6) | 4 (5)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 16 (28) | 6 (9)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 7 (50) | 44 (110) | 21 (145)
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 11 (12) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 19 (33) | 6 (7)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (10) | 7 (15) | 1 (15)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 9 (13) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (2) | 0 (0)
CSF protein increased (Investigations) | 1 (1) | 2 (3) | 4 (5)
Vitamin D decreased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (9) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 19 (24) | 14 (15)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Limb mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (2)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Amnesia (Nervous system disorders) | 1 (1) | 1 (3) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2)
Balance disorder (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4)
Cerebellar atrophy (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0)
Cerebral ventricle dilatation (Nervous system disorders) | 1 (1) | 4 (4) | 1 (2)
Coordination abnormal (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 8 (9) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (2) | 1 (2) | 1 (1)
Extensor plantar response (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 13 (25) | 6 (6)
Hypotonia (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Motor dysfunction (Nervous system disorders) | 1 (2) | 2 (3) | 0 (0)
Parkinsonism (Nervous system disorders) | 1 (2) | 0 (0) | 1 (3)
Pleocytosis (Nervous system disorders) | 1 (2) | 8 (16) | 2 (2)
Post-traumatic headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 6 (7)
Affect lability (Psychiatric disorders) | 1 (1) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 6 (6) | 7 (8)
Depressed mood (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (3)
Depression (Psychiatric disorders) | 1 (1) | 6 (6) | 4 (5)
Insomnia (Psychiatric disorders) | 1 (1) | 17 (17) | 6 (6)
Irritability (Psychiatric disorders) | 2 (3) | 4 (4) | 6 (8)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Haematoma (Vascular disorders) | 2 (2) | 1 (1) | 3 (4)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT03842969/Prot_SAP_000.pdf